CLINICAL TRIAL: NCT07241624
Title: Isometric Versus Isotonic Trunk Muscle Strength Training on Lung Function in Heavy Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Prof, MTI University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 31/7/2024-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Smokers

STUDY DESIGN:
Intervention Model Description: Single Blind ,RCT
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric Trunk Muscle Strength (Experimental): Participants will perform a series of isometric trunk exercises, such as planks and static bridges, three times a week
  Interventions: Other: Isometric trunk exercises
- Isotonic Trunk Muscle Strength (Experimental): Participants will engage in isotonic exercises, such as sit-ups and Russian twists, also three times a week.
  Interventions: Other: Isotonic trunk exercises
- Control (No Intervention): no intervention

INTERVENTIONS:
Other: Isometric trunk exercises — isometric trunk exercises, such as planks and static bridges, three times a week.
  Arms: Isometric Trunk Muscle Strength
Other: Isotonic trunk exercises — isotonic exercises, such as sit-ups and Russian twists, also three times a week.
  Arms: Isotonic Trunk Muscle Strength

SUMMARY:
Smoking is a major public health concern, significantly affecting lung function and overall respiratory health. Heavy smoking leads to chronic obstructive pulmonary disease (COPD), emphysema, and a decline in lung capacity. Exercise interventions, particularly those targeting the trunk muscles; have demonstrated potential in improving respiratory function. Trunk muscle strength is essential for optimal breathing mechanics, as these muscles support the chest wall and aid in the expansion and contraction of the lungs.

There are two primary types of muscle strength training: isometric and isotonic. Isometric exercises involve static contractions where the muscle length does not change, while isotonic exercises involve dynamic movements with muscle lengthening and shortening. Each type of training offers unique benefits and impacts on muscle strength and endurance. This proposal aims to compare the effects of isometric versus isotonic trunk muscle strength training on lung function among heavy smokers, providing insights into their relative efficacy in improving respiratory health. Thus, the objective of this study was to explore the therapeutic effectiveness of Isometric versus Isotonic Trunk Muscle Strength Training on Lung Function in Heavy Smokers.

DETAILED DESCRIPTION:
Smoking is the practice of inhaling and exhaling smoke from burning plant material, most commonly tobacco, which contains the addictive substance nicotine. It is a major public health concern and the leading preventable cause of death and disease, as it damages nearly every organ and significantly increases the risk for many conditions like various cancers, heart disease, stroke, and respiratory diseases such as COPD. Quitting smoking can reverse many of these effects.

Smoking has long been identified as a major risk factor for a variety of health issues, and its impact on physical fitness and muscle power is an area of growing concern. Trunk muscle power, which is crucial for maintaining posture, stability, and overall functional movement, can be significantly affected by smoking. The primary mechanism through which smoking influences trunk muscle power lies in its detrimental effects on cardiovascular health and respiratory function. Nicotine and other harmful substances in cigarettes reduce oxygen supply to muscles, impairing their ability to generate power efficiently. This reduction in oxygen availability not only affects muscle endurance but also increases fatigue, hindering the muscle's capacity to function effectively during physical activities.

Moreover, smoking contributes to systemic inflammation and oxidative stress, both of which can compromise muscle health. Chronic inflammation can lead to muscle wasting and weaken the structural integrity of muscle fibers, including those of the trunk muscles. Oxidative stress, resulting from an imbalance between the production of free radicals and the body's ability to counteract their harmful effects, accelerates muscle degradation and impairs muscle recovery post-exercise. This is particularly detrimental to trunk muscles, which are constantly engaged in stabilizing and supporting the body. The cumulative effect of these processes results in diminished muscle power and functional capacity, ultimately affecting an individual's quality of life and ability to perform daily activities.

In addition, smoking is often associated with a sedentary lifestyle, which further exacerbates the decline in trunk muscle power. Smokers may experience reduced motivation to engage in physical exercise due to decreased lung capacity and higher perceived exertion during activities. This lack of exercise contributes to muscle atrophy and a loss of muscle strength and power. Thus, the combination of smoking-induced physiological changes and lifestyle factors creates a cycle of declining muscle power. Addressing smoking cessation and promoting physical activity can therefore be vital strategies in preserving trunk muscle power and overall health, highlighting the importance of integrating health education and smoking cessation programs in health curricula.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20-45 years
* Self-reported heavy smokers (defined as smoking ≥20 cigarettes per day
* No participation in structured exercise programs in the past 6 months
* Capable of performing physical exercises

Exclusion Criteria:

* Diagnosed respiratory conditions other than smoking-related diseases (e.g., asthma)
* Cardiovascular diseases prohibiting physical exercise
* Recent surgeries or injuries affecting the trunk muscles
* Pregnant women

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) Moreover, smoking contributes to systemic inflammation and oxidative stress, both of which can compromise muscle health. Chronic inflammation can lead to muscle wasting and weaken the structural integrity of | at baseline after 8 weeks
  Forced Expiratory Volume in 1 second (FEV1) is a crucial measure of lung function that quantifies the volume of air a person can forcefully exhale in one second after a deep breath. It is used to assess the presence and severity of respiratory conditions
Forced Vital Capacity (FVC) | at base line after 8 weeks
  Forced Vital Capacity (FVC) is the maximum amount of air a person can forcibly exhale from the lungs after taking the deepest breath possible.
Peak Expiratory Flow (PEF) | at baseline and after 8 weeks
  Peak Expiratory Flow (PEF) is the maximum speed at which a person can exhale, providing a measure of airway obstruction in conditions like asthma. It's assessed using a peak flow meter to monitor respiratory health and guide treatment decisions.

SECONDARY OUTCOMES:
Trunk muscle strength | At baseline after 8 weeks
  Trunk muscle strength refers to the power and endurance of the core muscles, including the abdominal and lower back, which are essential for maintaining posture, stability, and efficient movement in daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt